CLINICAL TRIAL: NCT06106997
Title: Feasibility Study of an MRI-only Workflow: Use of Synthetic CTs Generated From MRI Data for MRI-based Radiotherapy
Brief Title: Clinical Feasibility of Brain Radiotherapy Using Synthetic CTs in an MRI-only Workflow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: sCT-Feasibility
Record Dates: First submitted 2023-10-16; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Brain Tumor, Primary; Brain Tumor - Metastatic
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sCT workflow (Other): sCT workflow
  Interventions: Radiation: brain radiotherapy

INTERVENTIONS:
Radiation: brain radiotherapy — brain radiotherapy planned on synthetic CTs

SUMMARY:
The goal of this observational study is to show the feasibility of an MRI-only workflow in brain radiotherapy. The main question it aims to answer is:

* Is an MRI-only workflow based on deep learning sCTs feasible in clinical routine? Participants will be treated as in clinical routine, but treatment planning will be based on sCTs, that are generated from MRI images. The dosimetrical equivalence to the standard CT based workflow will be tested at several points in the study.

DETAILED DESCRIPTION:
The purpose of this clinical study is to investigate the clinical feasibility of a deep learning-based MRI-only workflow for brain radiotherapy, that eliminates the registration uncertainty through calculation of a synthetic CT (sCT) from MRI data.

A total of 54 patients with an indication for radiation treatment of the brain and stereotactic mask immobilization will be recruited. All study patients will receive standard therapy and imaging including both CT and MRI. All patients will receive dedicated RT-MRI scans in treatment position. An sCT will be reconstructed from an acquired MRI DIXON-sequence using a commercially available deep learning solution on which subsequent radiotherapy planning will be performed. Through multiple quality assurance (QA) measures and reviews during the course of the study, the feasibility of an MRI-only workflow and comparative parameters between sCT and standard CT workflow will be investigated holistically. These QA measures include feasibility and quality of image guidance (IGRT) at the linear accelerator using sCT derived digitally reconstructed radiographs in addition to potential dosimetric deviations between the CT and sCT plan. The aim of this clinical study is to establish a brain MRI-only workflow as well as to identify risks and QA mechanisms to ensure a safe integration of deep learning-based sCT into radiotherapy planning and delivery.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patient older than 18 years
* Tumor or metastases in the brain
* Immobilization with stereotactic mask
* Treatment on stereotactic linear accelerator (2.5 mm leafs) equipped with 2D/2D X-ray system

Exclusion Criteria:

* Metal in the body, metal implants, pacemakers or other patient-specific factors that are a contraindication to an MRI scan
* Metal implants, pacemakers or other patient-specific factors associated with increased risk from an MRI scan
* Renal insufficiency (eGFR < 60 ml/min), allergy or other patient-specific factors that constitute a contraindication to contrast administration
* Renal insufficiency (eGFR < 60 ml/min), allergy or other patient-specific factors associated with an increased risk from contrast administration
* Patients who are institutionalized in care facilities, prisons or other supervised facilities.
* Patients under guardianship
* Non-consenting patients
* Pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that can successfully be treated in an MRI-only workflow | 12 month
  All criteria have to be met for the MRI-only workflow to be classified as successful:
  Verification criteria that will be assessed:
  1. Can the sCT be generated and is the sCT clinically utilizable?
  2. Are the three rotations needed for CT-MRI registration each ≤ 3°?
  3. Can a treatment plan be generated and verified using the sCT?
  4. Is the dosimetric difference between sCT and CT based treatment plan in the planning target volume ≤ 3%?
  5. Is the dosimetric difference between the sCT and CT based treatment plan in affected organs at risk (receiving > 10% of prescribed dose) ≤ 3%?
  6. Are the couch correction parameters during patient positioning in the rotational degrees of freedom ≤ 3°?

SECONDARY OUTCOMES:
Reasons that lead to unfeasibility of an MRI-only workflow | 12 month
  Presence (Yes/No) of individual reasons responsible for the unfeasibility of the MRI-only workflow, as assessed with a predefined checklist.
Dosimetric differences between MRI-only and standard workflow for radiotherapy treatment planning | 12 month
  Paired difference in Dose-volume-histogram parameters (Target coverage, mean, median, near maximum and minimum dose) between MRI-only and standard radiotherapy treatment workflow.
Measurement of intra-MRI patient positional changes | 12 month
  Patient shift (vector magnitude) and rotational errors occuring during the course of MRI acquisition due to patient movement, as assessed by rigid registration of the last acquired MRI sequence in reference to the first sequence.
Organ at risk contouring accuracy on MRI data | 12 month
  Similarity of organ at risk segmentations defined in MRI compared to reference segmentations defined in CT as assessed by the volumetric and surface Dice score, as well as mean surface and Hausdorff distances.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Bert, Prof. Dr. rer. nat, Principal Investigator — Universitätsklinikum Erlangen, Strahlenklinik; Florian Putz, PD Dr. med., Principal Investigator — Universitätsklinikum Erlangen, Strahlenklinik
Locations (1):
- Erlangen, Universitätsklinikum Strahlenklinik, Erlangen, Germany

REFERENCES:
- [Derived] Grigo J, Szkitsak J, Hofler D, Fietkau R, Putz F, Bert C. "sCT-Feasibility" - a feasibility study for deep learning-based MRI-only brain radiotherapy. Radiat Oncol. 2024 Mar 8;19(1):33. doi: 10.1186/s13014-024-02428-3. PMID 38459584